CLINICAL TRIAL: NCT05547607
Title: Observational Prospective Multicenter Study to Characterize the CLinical and DiagnoStiC FeAtures of Endocarditis in the ContemPorary Era
Brief Title: Clinical and Diagnostic Features of Endocarditis
Acronym: ENDO-LANDSCAPE
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Full Professor of Cardiology, University of Ferrara, University Hospital of Ferrara
Other Study IDs: 548/2022/Oss/AOUFe
Record Dates: First submitted 2022-09-09; First posted 2022-09-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- definite or high suspicion endocarditis: All consecutive patients referred for an echocardiography (transthoracic or transesophageal approach) with a high suspicion of endocarditis and those with a confirmed diagnosis of endocarditis independently by the request will be eligible for the study.
  Interventions: Diagnostic Test: advanced cardiac imaging
- negative examination with low suspicion of endocarditis: For patients with no evidence of endocarditis on their echocardiogram, data on the following will be collected: i) risk factors for endocarditis; i) size, type and position of valve prosthesis or other devices if present; iii) Duke criteria verification.
  Interventions: Diagnostic Test: advanced cardiac imaging

INTERVENTIONS:
Diagnostic Test: advanced cardiac imaging — In all patients with high suspected or confirmed endocarditis at the echocardiography the following information will be collected: 1) endocarditis risk factors, 2) type, size and position of infected valve or prosthesis, 3) echocardiographic data; 4) imaging technique used for diagnosis in addition to echocardiography; 5) management of the case performed by the endocarditis team (including cardiologist, microbiologist, cardiac surgeon, radiologist); 6) Duke criteria verification; 7) management of the case (conservative or invasive); 8) antibiotic therapy prescribed and timing; 9) follow-up at one year (death, cardiac surgery, stroke, re-infection).

SUMMARY:
The burden of endocarditis has changed in the last years due to an increase in percutaneous valve procedures offered to a more fragile, and old population. Therefore an update in epidemiology data is necessary. The Observational prospective multicenter study to characterize the cLinical ANd DiagnoStiC feAtures of endocarditis in the contemPorary Era, (ENDO-LANDSCAPE study) is an observational, multicenter and international study. The study has two arms: retrospective and prospective.

The retrospective arm will involve collecting data from patients discharged with a diagnosis of endocarditis between 2016 and 2022. The data obtained in the retrospective arm of the study will be utilized in a power calculation to determine the sample size for the prospective arm of the study. In the prospective phase in every participating center, all patients referred for echocardiography to assess for endocarditis and those with established endocarditis independent of the screened request will be eligible. Patients will then be stratified according to the presence or abscence of endocarditis. Those with an established diagnosis of endocarditis will be prospectively followed for outcomes.

DETAILED DESCRIPTION:
STUDY DESIGN The study will be multicenter and international with two arms: retrospective and prospective.

The retrospective arm will involve collecting data from patients discharged with a diagnosis of endocarditis between 2016 and 2022. The data obtained in the retrospective arm of the study will be utilized in a power calculation to determine the sample size for the prospective arm of the study.

Retrospective arm: It will be enrolled all patients discharged with a diagnosis of endocarditis. Data collected will be about: 1) position, size and type of valve or prosthesis infected, 2) echocardiographic data (both on transthoracic or transesophageal approach) regarding presence, size and morphology of vegetations and any other signs consistent with endocarditis (e.g.abscess, fistula, pseudoaneurysms), severity of valve disease; 3) imaging technique used for diagnosis in addition to echocardiography (computed tomography, positron emission computed tomography, single photon emission computed tomography); 4) management of the case performed by the endocarditis team (including cardiologist, microbiologist, cardiac surgeon, radiologist); 5) Duke criteria verification; 6) management of the case (conservative vs invasive); 7) antibiotic therapy prescribed and timing; 8) follow-up at one year (death, cardiac surgery, re-infection).

All data collected will be made anonymous. Data regarding follow-up will be obtained through medical chart or by hospital computer reporting systems. For this reason, a signed informed consent is not necessary for this phase of the study. All data will be collected in electronic format (e-CRF) on REDCAP.

Prospective arm: This phase will involve several international centres for a timeframe of 12 months.

All consecutive patients referred for a echocardiography with a suspicion of bacterial endocarditis and those with a confirmed diagnosis of endocarditis independently by the request will potentially be eligible for the study. Only the patients with a confirmed or with high suspicion of endocarditis will be prospectively followed for one year. As in the retrospective arm, these patients will be prospectively follow-up, and the following information collected: 1) type, size and position of infected valve or prosthesis, 2) echocardiographic data (both on transthoracic or transesophageal approaches) regarding presence, size and morphology of vegetations or other evidence of endocarditis (e.g. abscess, fistula, pseudoaneurysms), severity of valve disease; 3) imaging technique used for diagnosis in addition to echocardiography (computed tomography, positron emission computed tomography, single photon emission computed tomography); 4) management of the case performed by the endocarditis team (including cardiologist, microbiologist, cardiac surgeon, radiologist); 5) Duke criteria verification; 6) management of the case (conservative or invasive); 7) antibiotic therapy prescribed and timing; 8) follow-up at one year (death, cardiac surgery, re-infection).

For patients with no evidence of endocarditis on their echocardiogram, data on the following will be collected: i) size, type and position of valve prosthesis; ii) uke criteria verification.

In both cases a CRF will be filled. All patients enrolled in the prospective arm will sign a informed written consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years.
* all consecutive patients referred for echocardiography (transthoracic or transesophageal approach) to exclude endocarditis.
* patients with a diagnosis of endocarditis on echocardiography independently by the request for the exam.

Exclusion Criteria:

* patient's refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred for a echocardiography with a suspicion of bacterial endocarditis and those with a confirmed diagnosis of endocarditis independently by the request will potentially be eligible for the study. Only the patients with a positive findings of endocarditis will be prospectively followed for one year. For patients with no evidence of endocarditis on their echocardiogram, data on the following will be collected: i) size, type and position of valve prosthesis; ii) Duke criteria verification.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
incidence of endocarditis | 1 year
  the incidence of endocarditis in patients with native valve, surgical implanted prosthesis, percutaneously corrected valve disease, other devices

SECONDARY OUTCOMES:
Appropriateness of requests for echocardiography to exclude endocarditis | day 1
  The investigator will asses based on clinical and laboratory data if the suspicion of endocarditis was reliable and then the request of echocardiography appropriate
All-cause mortality of surgically treated endocarditis | 1 year
  All-cause mortality of surgically treated endocarditis
All-cause mortality of medically managed endocarditis | 1 year
  All-cause mortality of medically managed endocarditis
Cerebrovascular accident | 1 year
  Cumulative occurrence of ischemic stroke and transient ischemic attack
Re-infection in invasively treated endocarditis | 1 year
  Cumulative occurrence of new hospitalization for endocarditis (or other infection related to the surgical intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Pavasini, MD, Principal Investigator — University Hospital of Ferrara
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request

REFERENCES:
- [Derived] Pavasini R, Sinning C, Campo G, Tan TC. ObsErvatioNal prospective multicenter stuDy tO characterize the cLinical ANd DiagnoStiC feAtures of endocarditis in the contemPorary Era (ENDO-LANDSCAPE study): rationale and design. J Cardiovasc Med (Hagerstown). 2023 Jun 1;24(6):354-360. doi: 10.2459/JCM.0000000000001469. Epub 2023 Apr 6. PMID 37021952